CLINICAL TRIAL: NCT02879552
Title: Tarsal Platform Show After Upper Eyelid Blepharoplasty With or Without Brassiere Sutures
Brief Title: TPS After Upper Blepharoplasty
Status: Completed | Type: Observational
Sponsor: Instituto de Olhos de Goiania (Other)
Collaborators: Centro de Referência em Oftalmologia (Unknown)
Responsible Party: Sponsor
Other Study IDs: MR-01-2016
Record Dates: First submitted 2016-08-21; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Efficacy of a Technique (Brassiere Sutures)
Keywords: Upper blepharoplasty; brassiere sutures; tarsal platform show; eyeshadow space; brow fat span
MeSH Terms: interventions — Blepharoplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Traditional upper blepharoplasty: Patients with an odd total number of letters in their first name received traditional upper blepharoplasty.
  Interventions: Procedure: Brassiere suture with blepharoplasty
- Brassiere suture with blepharoplasty: The rest of the patients received orbicularis oculi muscle fixation to periosteum (brassiere sutures)
  Interventions: Procedure: Traditional upper blepharoplasty

INTERVENTIONS:
Procedure: Traditional upper blepharoplasty — The skin incisions were marked using a skin marking pen. Preseptal orbicularis skin and muscle were removed using a size-15 scalpel blade and scissors. Hemostasis was achieved with conservative electrocuatery. The skin was closed with a running 6-0 nylon suture.
  Groups: Brassiere suture with blepharoplasty
Procedure: Brassiere suture with blepharoplasty — Prior to skin closure as above, three 6-0 polyglactin sutures are passed along the lateral fourth of the orbital rim. The sutures attach the inferior orbicularis oculi edge to the arcus marginalis of lateral ROOF. Sutures are placed until there is a visible "plumping" of the sub-brow tissues.
  Groups: Traditional upper blepharoplasty

SUMMARY:
Increased tarsal platform show (TPS) and decreased brow fat span (BFS) are associated with favorable results in women undergoing cosmetic blepharoplasty. The authors evaluate the efficacy of a technique (brassiere sutures) to increase TPS and decrease the BFS.

DETAILED DESCRIPTION:
This is a prospective, randomized, comparative, case series study of 100 eyelids (50 consecutive women patients) treated with cosmetic upper blepharoplasty by a single surgeon. Patients were randomized to receive traditional upper blepharoplasty with a single running suture skin closure versus orbicularis oculi muscle fixation to periosteum (brassiere sutures) prior to skin closure. Patient age, follow-up length, complications and treatment were analyzed. The mean of TPS, BFS and TPS/BFS ratio was measured before and after surgery at 3 anatomic landmarks.

56 eyelids (28 patients) were treated with traditional single suture blepharoplasty and 44 eyelids (22 patients) had brassiere sutures. After surgery, the mean change in TPS was 2.10 mm with brassiere sutures compared to 2.04 mm without (p <.001). The mean change in BFS was 3.33 mm with brassiere sutures compared to 3.19 mm without (p <.001), The mean change in TPS:BFS ratio at all 3 anatomic landmarks was statistically significant in both groups but the change was statistically greater with the use of brassiere sutures (p <.001).

Brassiere sutures during upper blepharoplasty were associated with a postoperative increase in TPS decrease in BFS, and increase in TPS/BFS.

ELIGIBILITY:
Inclusion Criteria:

* Female underwent cosmetic upper blepharoplasty and brassiere suture with blepharoplasty

Exclusion Criteria:

* History of thyroid eye disease, levator dehiscence ptosis, blepharospasm, facial nerve paresis, a history of previous upper facial surgery or trauma, and postoperative follow-up for less than 6 months.

Ages: 35 Years to 81 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective, randomized, observational case series study included 110 eyelids (50 patients) that underwent cosmetic upper blepharoplasty and brassiere suture.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Eyelid measurements of traditional blepharoplasty and brassiere suture, before and after surgery | 6 months

SECONDARY OUTCOMES:
Asymmetry of TPS and BFS in traditional blepharoplasty and brassiere suture | 6 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Figueiredo MN, Tao J, Akaishi P, Limongi RM. Tarsal platform show after upper eyelid blepharoplasty with or without brassiere sutures. Arq Bras Oftalmol. 2017 Nov-Dec;80(6):345-349. doi: 10.5935/0004-2749.20170085. PMID 29267567